CLINICAL TRIAL: NCT06420180
Title: The Effect of Lower Limb Rotation on Clinical Outcomes After Arthroscopic Management in Patients With Symptomatic Femoroacetabular Impingement Syndrome
Brief Title: Effect of Lower Limb Rotation on Clinical Outcomes After Arthroscopic Management in Patients With Symptomatic Femoroacetabular Impingement Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, mahmoud ahmed awad elmetwally, Assistant Lecturer of Orthopedic Surgery, Al-Azhar University
Other Study IDs: lower limb rotation on FAI
Record Dates: First submitted 2024-05-11; First posted 2024-05-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Femoro Acetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hip arthroscopy — CT rotational profile Will be used for measurement of LL rotational abnormality.
  MRI will be evaluated for the presence of labral tears, chondral lesions, ligamentum teres pathology, and other soft-tissue disorders.
  Other Names: MRI; CT

SUMMARY:
To determine

* The prevalence of abnormalities of femoral and acetabular versions and tibial torsion in symptomatic (FAI) Syndrome.
* Analyse the subgroups of specific hip pathomorphologies associated with rotational abnormalities of lower limb (LL).
* Which specific hip subtypes of (FAI) are associated with rotational abnormalities,
* Outcomes of arthroscopic treatment of (FAI) syndrome in patients with rotational abnormalities compared with a control group of patients with normal rotation.

DETAILED DESCRIPTION:
Femoroacetabular impingement (FAI) is characterised by an abnormal contact between the acetabulum and the femur, limiting range of motion and leading to hip pain and disability.

(FAI) can be classified into three categories according to the specific pathomorphology involved. Cam type (FAI) represents asphericity of the femoral head due to abnormal morphology at the head neck junction. Pincer-type (FAI) on the other hand, occurs due to over-coverage of the femoral head by the acetabulum and premature contact between the acetabulum and femoral neck. Some patients may present with both of these abnormalities, known as mixed-typed (FAI).

There is an interest in the role of acetabular and femoral versions and tibial torsion in (FAI). Lerch et al. found that 68% of 538 hips presenting with (FAI) or dysplasia showed abnormal femoral and/or acetabular versions. A more recent study by Lerch et al. also found abnormal tibial torsion in 42% of patients with (FAI) and dysplasia. It has been further speculated that excessive femoral anteversion or femoral retroversion may also play a role in the pathogenesis and treatment of (FAI). Excessive femoral retroversion has been considered by some to be a relative contraindication to corrective (FAI) surgery, as it has been found to be a risk factor for poor outcomes after hip arthroscopy for (FAI). Similarly, increased femoral version is a risk factor for inferior clinical outcomes after hip arthroscopy. Abnormalities of femoral version and tibial torsion were associated with anterior knee pain, knee osteoarthritis, and patellar instability. But the influence of combined abnormalities of femoral version and tibial torsion (combined torsional malalignment) for patients with hip pain is unknown.

So, investigator hypothesized that patients with symptomatic (FAI) display significant rotation abnormalities of the acetabulum or femur and tibial and that the rotational abnormalities would portend an inferior prognosis when compared with a pair-matched control group of patients with normal range of lower limb rotation and patients with significant rotational abnormalities would have differing intraoperative hip pathology.

ELIGIBILITY:
Inclusion Criteria:

* • Accepted to participate in the study (signing informed consent).

  * Skeletal maturity (Risser V score).
  * If their radiographic imaging, history, and physical examination demonstrated evidence of FAI or labral tears; if they experienced moderate to severe pain that was unresponsive to at least 3 months of nonsurgical treatment, including physical therapy, nonsteroidal anti-inflammatory drugs, and activity modification

Exclusion Criteria:

* • Incomplete radiographic documentation.

  * Previous surgery of the acetabulum, femur and/or tibia altering their version.
  * Skeletally immature hips (stage IV according to Risser).
  * Posttraumatic conditions.
  * If they were previously diagnosed with an ipsilateral hip condition, such as avascular necrosis, legg-calvé-perthes disease, or slipped capital femoral epiphysis.
  * If their tönnis grade of osteoarthritis is >1.
  * Hip dysplasia will be defined as a lateral centre-edge angle (LCEA) less than 22°.
  * Patients with rheumatologic diseases.
  * Patients at risk of radiation exposure, such as pregnant women and patients after neoplastic diseases.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: study will be conducted on patient aged between 18 to 45 years with radiographic imaging, history, and physical examination demonstrated evidence of FAI or labral tears; if they experienced moderate to severe pain that was unresponsive to at least 3 months of nonsurgical treatment, including physical therapy, nonsteroidal anti-inflammatory drugs, and activity modification
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
prevalence of lower limb rotation in FAI | baseline
  determine the prevalence of abnormalities of femoral and acetabular versions and tibial torsion in symptomatic FAI Syndrome.
2 years outcome of arthroscopic treatment of 50 patients with FAI syndrome using modified Harris Hip Score (mHHS). | 2 years
  determine Outcomes of arthroscopic treatment of FAI syndrome in patients with rotational abnormalities compared with patients with normal rotation.
  normal rotation according to preoperative CT rotational profile: Acetabular version angle between 10⁰ to 25⁰. Femoral version angle between 10⁰ to 25⁰. Tibial torsion angle between 25⁰ to 40⁰. clinical outcome of arthroscopic treatment of patients with FAI syndrome using modified Harris Hip Score (mHHS) will be done preoperatively and postoperatively at 1.5 months, 3 months, 6 months, 1 year, and 2 years.
  The modified Harris hip score (mHHS) will be scored from 0 (worst functional outcome and maximum pain) to 100 points (best functional outcome and least pain)
2 years outcome of arthroscopic treatment of 50 patients with FAI syndrome using Nonarthritic Hip Score (NAHS). | 2 years
  determine Outcomes of arthroscopic treatment of FAI syndrome in patients with rotational abnormalities compared with patients with normal rotation.
  normal rotation according to preoperative CT rotational profile: Acetabular version angle between 10⁰ to 25⁰. Femoral version angle between 10⁰ to 25⁰. Tibial torsion angle between 25⁰ to 40⁰. clinical outcome of arthroscopic treatment of patients with FAI syndrome using Nonarthritic Hip Score (NAHS) will be done preoperatively and postoperatively at 1.5 months, 3 months, 6 months, 1 year, and 2 years.
  This score is divided into four domains: pain, mechanical symptoms, physical function, and level of activity.
  The maximum score is 100 indicating normal hip function.
2 years outcome of arthroscopic treatment of 50 patients with FAI syndrome using Hip Outcome Score-Sports Specific Subscale (HOS-SSS) | 2 years
  determine Outcomes of arthroscopic treatment of FAI syndrome in patients with rotational abnormalities compared with patients with normal rotation.
  normal rotation according to preoperative CT rotational profile: Acetabular version angle between 10⁰ to 25⁰. Femoral version angle between 10⁰ to 25⁰. Tibial torsion angle between 25⁰ to 40⁰. clinical outcome of arthroscopic treatment of patients with FAI syndrome using Hip Outcome Score-Sports Specific Subscale (HOS-SSS) will be done preoperatively and postoperatively at 1.5 months, 3 months, 6 months, 1 year, and 2 years.
  The (HOS-SSS) is a patient-completed measure that consists of "(9 scored items) in which the response options are presented as 5-point Likert scales. Scores for each subscale range from 0% (least function) to 100% (most function).

REFERENCES:
- [Background] Arshad Z, Maughan HD, Sunil Kumar KH, Pettit M, Arora A, Khanduja V. Over one third of patients with symptomatic femoroacetabular impingement display femoral or acetabular version abnormalities. Knee Surg Sports Traumatol Arthrosc. 2021 Sep;29(9):2825-2836. doi: 10.1007/s00167-021-06643-3. Epub 2021 Jul 6. PMID 34228156
- [Background] Lerch TD, Todorski IAS, Steppacher SD, Schmaranzer F, Werlen SF, Siebenrock KA, Tannast M. Prevalence of Femoral and Acetabular Version Abnormalities in Patients With Symptomatic Hip Disease: A Controlled Study of 538 Hips. Am J Sports Med. 2018 Jan;46(1):122-134. doi: 10.1177/0363546517726983. Epub 2017 Sep 22. PMID 28937786
- [Background] Lerch TD, Liechti EF, Todorski IAS, Schmaranzer F, Steppacher SD, Siebenrock KA, Tannast M, Klenke FM. Prevalence of combined abnormalities of tibial and femoral torsion in patients with symptomatic hip dysplasia and femoroacetabular impingement. Bone Joint J. 2020 Dec;102-B(12):1636-1645. doi: 10.1302/0301-620X.102B12.BJJ-2020-0460.R1. PMID 33249913
- [Background] Imhoff FB, Funke V, Muench LN, Sauter A, Englmaier M, Woertler K, Imhoff AB, Feucht MJ. The complexity of bony malalignment in patellofemoral disorders: femoral and tibial torsion, trochlear dysplasia, TT-TG distance, and frontal mechanical axis correlate with each other. Knee Surg Sports Traumatol Arthrosc. 2020 Mar;28(3):897-904. doi: 10.1007/s00167-019-05542-y. Epub 2019 May 24. PMID 31127313
- [Background] Grunwald L, Histing T, Springer F, Keller G. MRI-based torsion measurement of the lower limb is a reliable and valid alternative for CT measurement: a prospective study. Knee Surg Sports Traumatol Arthrosc. 2023 Nov;31(11):4903-4909. doi: 10.1007/s00167-023-07533-6. Epub 2023 Aug 17. PMID 37589766
- [Background] Suarez-Ahedo C, Gui C, Rabe SM, Chandrasekaran S, Lodhia P, Domb BG. Acetabular Chondral Lesions in Hip Arthroscopy: Relationships Between Grade, Topography, and Demographics. Am J Sports Med. 2017 Sep;45(11):2501-2506. doi: 10.1177/0363546517708192. Epub 2017 Jun 7. PMID 28590784